CLINICAL TRIAL: NCT05529459
Title: ASSIST Trial Anatomic Versus Physiologic Guidance for Complete Revascularization With Drug Eluting Stent Implantation in Patients With Coronary Artery Disease
Brief Title: Anatomic Versus Physiologic Guidance for Complete Revascularization With DES Eluting in Patients With CAD
Acronym: ASSIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seung-Whan Lee, M.D., Ph.D. (Other)
Collaborators: Biotronik Korea Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Seung-Whan Lee, M.D., Ph.D., Principal investigator, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022-1298
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- quantitative coronary angiography-guided percutaneous coronary intervention (Experimental): Successful revascularization of all coronary artery lesions or segments ≥2.25 mm* in diameter with ≥50% diameter stenosis by QCA regardless of their functional significance
  Interventions: Procedure: Percutaneous Coronary Intervention
- fractional flow reserve-guided PCI (Active Comparator): Successful revascularization of all coronary artery lesions or segments ≥2.25 mm in diameter with evidence of ischemia or hemodynamic significance by FFR ≤ 0.80 regardless of their anatomic severity†
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Percutaneous Coronary Intervention

SUMMARY:
This study is to compare clinical outcomes between quantitative coronary angiography-guided anatomic complete revascularization and fractional flow reserve-guided physiologic complete revascularization in patients with significant coronary artery disease undergoing percutaneous coronary intervention with drug eluting stent

DETAILED DESCRIPTION:
This is a prospective, multicenter center, open-label, randomized trial to compare QCA-guided versus FFR-guided CR strategies in patients with significant CAD who are undergoing PCI with DES. Patients with symptoms or evidence of myocardial ischemia are eligible for enrollment if there have stenotic lesions with a diameter stenosis of 50%-90% in major epicardial coronary arteries ≥ 2.25 mm in diameter by visual estimation, and CR is expected to be achievable by PCI. The detailed information for inclusion and exclusion criteria is described below in the session 4. Patients meeting inclusion criteria without any exclusion criteria will be randomized to either QCA-guided CR or FFR-guided CR group. In the QCA-guided CR group, PCI will be performed if there are lesions with diameter stenosis ≥ 50% by QCA during the index procedure (and, if necessary, planned staged procedure). In the FFR-guided CR group, FFR is measured for the target coronary lesions, and then PCI will be performed for the lesions with FFR ≤0.80. Post-PCI FFR measurement is strongly recommended. However, additional procedures are not recommended based on post-PCI FFR value because there is no consensus of the optimal cut-off value to define physiologic CR. In both QCA-guided and FFR-guided PCI groups, imaging guidance during PCI is left at the discretion of the operator. However, routine high pressure post-dilation with noncompliant balloons is recommended to achieve optimal stent expansion with minimal residual stenosis (diameter stenosis < 10% on visual estimation). Patients will be followed clinically at 1, 6, 12 months, and then upto 5 years after the index procedure

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 19and older
* Typical chest pain or objective evidence of myocardial ischemia suitable for PCI Significant lesions with a diameter stenosis of 50-90% in major epicardial coronary arteries ≥ 2.25 mm in diameter by visual estimation.
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Coronary lesions resulting in the expected inability to perform FFR (ex, severe tortuosity or extreme angulation of the vessels)
* Chronic total occlusion
* Failed PCI of severe stenotic (diameter stenosis > 90%) or ACS culprit lesions
* Previous PCI within 6 months before the index procedure
* Previous coronary artery bypass graft surgery
* Cardiogenic shock or hemodynamic instability
* Left ventricular dysfunction (ejection fraction < 35%)
* Life expectancy < 1 years for any non-cardiac or cardiac causes
* Any surgery requiring general anesthesia or discontinuation of aspirin and/or an ADP antagonist is planned within 12 months after the procedure
* A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer
* Patient's pregnant or breast-feeding or child-bearing potential.
* A known intolerance to antiplatelet agents (aspirin, clopidogrel, prasugrel or ticagrelor)
* Hypersensitivity or contraindication to DES material and its degradants and cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers that cannot be adequately pre-medicated
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the investigator, would preclude safe completion of the study
* Unwillingness or inability to comply with the procedures described in this protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with death | 12month
  Major adverse cardiac events are defined as all-cause death
Number of Participants with MI | 12month
  Non-fatal myocardial infarction includes both spontaneous MI and periprocedural MI.
Number of Participants with unplanned repeat revascularization | 12month
  Unplanned repeat revascularization is defined as revascularization of any diseased coronary arteries ≥ 2.0 mm in diameter by QCA due to recurred angina with at least one of the following: (1) positive non-invasive test, (2) positive invasive physiologic test, or (3) presence of diameter stenosis ≥50% by QCA.

SECONDARY OUTCOMES:
Number of Participants with death | 5years
  Major adverse cardiac events are defined as all-cause death
Number of Participants with MI | 5years
  Non-fatal myocardial infarction includes both spontaneous MI and periprocedural MI.
Number of Participants with unplanned repeat revascularization | 5years
  Unplanned repeat revascularization is defined as revascularization of any diseased coronary arteries ≥ 2.0 mm in diameter by QCA due to recurred angina with at least one of the following: (1) positive non-invasive test, (2) positive invasive physiologic test, or (3) presence of diameter stenosis ≥50% by QCA.
Number of Participants with bleeding | 5years
  Major or minor bleeding according to definitions from TIMI
Number of Participants with rehospitalization | 5years
  Rehospitalization for an acute coronary syndrome or repeat PCI
Self-rated health on a vertical visual analogue scale by EQ5D | 5years
  EQ-5D is a standardized measure of health-related quality of life developed by the EuroQol Group and provides a simple and general questionnaire for use in clinical assessments
cost-effectiveness | 5years
  Procedure-related cost during index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Whan Lee, Investigator, Principal Investigator — Asan Medical Center
Locations (17):
- South Korea (17):
  - Hallym University Sacred Heart Hospital, Anyang
  - Bucheon Sejong Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Chungbuk National University Hospital, Cheongju-si
  - Daegu Veterans Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Gangneung Asan Hospital, Gangneung
  - Wonkwang University Hospital, Iksan
  - Kwangju Christian Hospital, Kwangju
  - Inje University Pusan Paik Hospital, Pusan
  - Bundang CHA Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Veterans Hospital Service Medical Center, Seoul
  - The Catholic University of Korea, ST. Vincent's Hospital, Suwon
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No